CLINICAL TRIAL: NCT03668301
Title: Differences Between Central Venous and Cerebral Tissue Oxygen Saturation in Anesthetized Patients With Diabetes Mellitus
Brief Title: Cerebral-tissue Oxygen Balance Affected by Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Collaborators: Hungarian Basic Research Council (Other)
Responsible Party: Principal Investigator, Barna Babik, Principal Investigator, Senior lecturer, Szeged University
Other Study IDs: WHO2788
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus (D003920); Cardiac Surgical Procedures (D006348); Near-Infrared (D019265)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group CPB-T2DM: Patients with diabetes mellitus undergoing cardiac surgery with cardiopulmonary bypass
- Group OPCAB-T2DM: Patients with diabetes mellitus undergoing cardiac surgery without cardiopulmonary bypass
- Group CPB-C: Control patients undergoing cardiac surgery with cardiopulmonary bypass
- Group OPCAB-C: Control patients undergoing cardiac surgery without cardiopulmonary bypass

SUMMARY:
The brain has high oxygen extraction, thus the regional cerebral tissue oxygen saturation (rSO2) is lower than the central venous oxygen saturation (ScvO2). The investigators hypothesized that diabetes widens the physiological saturation gap between ScvO2 and rSO2 (gSO2), and the width of this gap may vary during various phases of cardiac surgery. The investigators involve cardiac surgery patients with and without type 2 diabetes mellitus (T2DM) undergoing either off-pump coronary artery bypass (OPCAB) or other cardiac surgery necessitating cardiopulmonary bypass (CPB). rSO2 is measured by near-infrared spectroscopy (NIRS) and ScvO2 is determined simultaneously from central venous blood. rSO2 is registered before and after anesthesia induction and at different stages of the surgery.

DETAILED DESCRIPTION:
One hour before the surgery, patients are premedicated with lorazepam (per os, 2.5 mg). Before induction of anesthesia, the NIRS sensors (INVOS 3100, Somanetics, MI, USA) arepositioned on both sides of the forehead. Sensors to detect depth of anesthesia are also mounted on the forehead to monitor EMG and EEG activities. These signals are used to calculate response (RE) and state entropy (SE), respectively (GE Healthcare, Chicago, USA). Induction of anesthesia is achieved by iv midazolam (30 μg/kg), sufentanil (0.4-0.5 μg/kg), and propofol (0.3-0.5 mg/kg), and iv propofol (50 mg/kg/min) is administered to maintain anesthesia. Intravenous boluses of rocuronium (0.6 mg/kg for induction and 0.2 mg/kg every 30 minutes for maintenance) is administered iv to ensure neuromuscular blockade. A cuffed tracheal tube (internal diameter of 7, 8, or 9 mm) is used for tracheal intubation, and patients are mechanically ventilated (Dräger Zeus, Lübeck, Germany) in volume-controlled mode with decelerating flow. A tidal volume of 7 ml/kg and a positive end-expiratory pressure of 4 cmH2O are applied, and the ventilation frequency is adjusted to 12-14 breaths/min to maintain end-tidal CO2 partial pressure of 36 38 mmHg. Mechanical ventilation is performed with a fraction of inspired oxygen of 0.5 during the entire OPCAB procedure and before CPB, and it is increased to 0.8 after CPB. As a standard part of the cardiac anesthesia procedure, esophageal and rectal temperature probes are introduced, and a central venous line is inserted into the right jugular vein. The left radial artery is also cannulated to monitor systolic, diastolic and mean arterial (MAP) blood pressures and arterial blood gas samples.

The membrane oxygenator is primed with 1,500 ml lactated Ringer's solution prior to CPB. Intravenous heparin (150 or 300 U/kg for OPCAB and CPB procedures, respectively) is injected into the patient, and an activated clotting time of 300 s is achieved during OPCAB and of 400 s during CPB procedures. During CPB, mild hypothermia is allowed, the mechanical ventilation is stopped, and the ventilator is disconnected without applying positive airway pressure. Before restoring ventilation, the lungs are inflated 3-5 times to a peak airway pressure of 30 cmH2O to facilitate lung recruitment. Normothermia is maintained in the OPCAB patients.

After securing arterial and peripheral venous lines and placement of NIRS and entropy sensors, data collection is initiated immediately before anesthesia induction in all groups of patients. Since catheterization of the jugular vein is scheduled after anesthesia induction, ScvO2 and gSO2 data are not available at the first protocol stage. After induction and before surgical incision, all measurements are repeated. For the patients undergoing CPB procedures, the whole data set is registered at the beginning of CPB after clamping the aorta and 5 min before the end of CPB. For the patients undergoing OPCAB procedures, collection of the full set of data is performed during performance of the first proximal anastomosis between the aorta and saphenous vein graft. The final stage of the protocol is allocated to the end of the operation after sternal closure. All invasive (i.e. arterial and venous blood gas) and non-invasive (i.e. NIRS) data are registered simultaneously at each protocol stage.

Sample sizes are estimated to enable the detection of a 10% difference in the primary outcome parameter gSO2 that we considered clinically significant. Accordingly, sample-size estimation based on an ANOVA test with four groups of patients indicated that 24 patients were required in each group to detect a significant difference between the protocol groups (the assumed variability of 10%, power of 80% and the significance level of 5%).

Two-way repeated measures ANOVA with the inclusion of an interaction term is used for all measured variables with the protocol stage as within-subject factor (protocol stages) and group allocation as between-subject factor to establish the effects of T2DM and the surgical procedure on the oxygen saturation indices.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with or without diabetes mellitus,
* Age between 18-80 years

Exclusion Criteria:

* Patients older than 80 years of age,
* Poor ejection fraction (<40%),
* Unilateral internal carotid stenosis (>75%),
* Medical history of smoking,
* Medical history of chronic obstructive pulmonary disease
* Medical history of stroke

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients enrolled at the Second Department of Internal Medicine and Cardiology Center Cardiac Surgical Unit, University of Szeged
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation | Intraoperative interval during cardiac surgery starting from anesthsia induction until end of the surgery.
  The spatially resolved continuous-wave NIRS technique is applied to estimate cerebral tissue oxygen saturation. This monitor uses two different wavelengths (730 and 810 nm) and has two detectors positioned 3 and 4 cm from the light source. Computing the differences between the intensity of the emitted and the reflected light 13 with two receivers 14 allows the measurement of the oxygen saturation of the cerebral cortex. In this study, two adult sensors are applied on the left and right sides of the patient's forehead symmetrically, and the cerebral-tissue oxygen saturation is monitored continuously during the surgical procedures and the data are registered in each protocol stage. The mean value of the rSO2 measured by the sensors is calculated for each protocol stage and used for further analyses.
Central venous oxygen saturation | Intraoperative interval during cardiac surgery starting from anesthsia induction until end of the surgery.
  The central venous oxygen saturation is measured from central venous blood samples (Radiometer ABL 505, Copenhagen, Denmark). The proper positioning of the central venous catheter is verified by the surgeon via manually palpating the catheter tip.